CLINICAL TRIAL: NCT03796286
Title: A Randomized, Crossover Study to Assess the Effects of Dietary Fiber-containing Bars on Postprandial Glucose and Insulin Responses.
Brief Title: A Randomized, Crossover Study to Assess the Effects of Dietary Fiber-containing Bars on Glucose and Insulin Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Center for Metabolic and Cardiovascular Research (Other)
Collaborators: Ingredion Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: MB-1805
Record Dates: First submitted 2019-01-04; First posted 2019-01-08 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Blood Glucose; Insulin Sensitivity; Dietary Fiber
Keywords: Postprandial glucose; Meal tolerance test
MeSH Terms: conditions — Insulin Resistance | interventions — Dietary Fiber

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, three-treatment, crossover trial with one screening/baseline visit and three test visits. At each testing visit, the study product (a bar) will be consumed with water.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study site will be provided pre-packaged, sealed containers of control (a bar with no fiber) and active study products (a bar with 10 grams of fiber and a bar with 20 grams of fiber). Each product container will be labeled with the lot number, expiration date, and blinded product code.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control bar (0 g fiber) (Placebo Comparator): Each subject will be randomly assigned to consume a control sports bar-type product (0 grams of fiber) at one treatment visit.
  Interventions: Other: Control bar (0 g fiber)
- Medium-fiber bar (Experimental): Each subject will be randomly assigned to consume sports bar-type product (containing 10 grams of fiber) at one treatment visit.
  Interventions: Other: Medium-fiber bar
- High-fiber bar (Experimental): Each subject will be randomly assigned to consume sports bar-type product (containing 20 grams of fiber) at one treatment visit.
  Interventions: Other: High-fiber bar

INTERVENTIONS:
Other: Medium-fiber bar — Each subject will receive one control and two active treatments in a crossover design. The two active treatments are dietary fiber-containing bars at two doses of fiber. The control bar will not contain fiber.
  Arms: Medium-fiber bar
Other: High-fiber bar — Each subject will receive one control and two active treatments in a crossover design. The two active treatments are dietary fiber-containing bars at two doses of fiber. The control bar will not contain fiber.
  Arms: High-fiber bar
Other: Control bar (0 g fiber) — Each subject will receive one control and two active treatments in a crossover design. The two active treatments are dietary fiber-containing bars at two doses of fiber. The control bar will not contain fiber.
  Arms: Control bar (0 g fiber)

SUMMARY:
This randomized, crossover study will include four clinic visits: one screening (day -7) and three test visits (days 0, 2, 4). The objective of this study is to assess the effects of dietary fiber-containing bars, at two doses of fiber, compared to a control product, on postprandial glucose and insulin responses in healthy adult men and women.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18-65 y of age, inclusive.
* Subject has a body mass index of 18.5 to 32.0 kg/m, inclusive.
* Subject is judged by the Investigator to be in generally good health on the basis of medical history and screening measurements.
* Subject is willing to consume the study products as described in the protocol.
* Subject is willing to maintain usual diet and activity patterns throughout the study.
* Subject has no plans to change smoking or other nicotine use during the study period.
* Subject is willing and able to attend all clinic visits.
* Subject has a vein access scale score of 7-10.
* Subject understands the study procedures and signs forms documenting informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator and is willing to complete study procedures.

Exclusion Criteria:

* Individual has a clinically significant gastrointestinal, endocrine (including Type 1 and Type 2 diabetes mellitus), cardiovascular, renal, hepatic, pulmonary, pancreatic, neurologic, or biliary disorder.
* Subject has pre-diabetes (fasting capillary glucose between 100 and 125 mg/dL) at screening. One re-test on a separate day will be allowed for subjects with no known history of pre-diabetes or diabetes who have a capillary glucose of 100 - 110 mg/dL at screening (visit 1).
* Individual has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg) at screening.
* Individual has a history of cancer in the prior 2 years, except for non-melanoma skin cancer.
* Individual has extreme dietary habits (e.g., Atkins, vegan).
* Individual has had weight change of ±4.5 kg (10 lbs) in the previous 3 months.
* Individual has a known allergy, sensitivity, or intolerance to any ingredients in the study products.
* Individual is a female, who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period.
* Individual has been exposed to any non-registered drug product within 30 days of screening.
* Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent or comply with the study protocol, or which might confound the interpretation of the study results or put the person at undue risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2019-02-27 (Actual); Study Completion 2019-02-27 (Actual)

PRIMARY OUTCOMES:
Change in the incremental area under the curve for capillary glucose. | Up to 120 minutes - measured at each treatment visit
  Differences between the dietary fiber and control conditions following a breakfast meal tolerance test (MTT) completed at visits 2, 3, and 4 in the incremental AUC (iAUC) from pre-breakfast intake to 2 hours post breakfast intake for capillary glucose.

SECONDARY OUTCOMES:
Change in the incremental area under the curve for venous glucose. | Up to 120 minutes - measured at each treatment visit
  Differences between the dietary fiber and control conditions following a breakfast meal tolerance test (MTT) completed at visits 2, 3, and 4 in the incremental AUC (iAUC) from pre-breakfast intake to 2 hours post breakfast intake for venous glucose.
Change in the incremental area under the curve for venous insulin. | Differences between the dietary fiber and control conditions following a breakfast meal tolerance test (MTT) completed at visits 2, 3, and 4 in the incremental AUC (iAUC) from pre-breakfast intake to 2 hours post breakfast intake for venous glucose.
  Differences between the dietary fiber and control conditions following a breakfast meal tolerance test (MTT) completed at visits 2, 3, and 4 in the incremental AUC (iAUC) from pre-breakfast intake to 2 hours post breakfast intake for venous insulin.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Maki, PhD, Study Director — MB Clinical Research and Consulting LLC
Locations (2):
- United States (2):
  - MB Clinical Research, Boca Raton, Florida
  - Great Lakes Clinical Trials, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No